CLINICAL TRIAL: NCT05967780
Title: Comparison of Open Heart Surgery Patients With Forward Head Posture With and Without Perioperative Therapeutic Exercise on Craniovertebral Angle, Pulmonary Function, Balance and Quality of Life
Brief Title: Comparison of Open Heart Surgery Patients With Forward Head Posture With and Without Perioperative Therapeutic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.TUMS.FNM.REC.1402.060
Record Dates: First submitted 2023-07-04; First posted 2023-08-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Rehabilitation
Keywords: Balance; Craniovertebral angle; Forward head posture; Open heart surgery; Pulmonary function; Quality of life; Strengthening; Stretching
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Patients with FHP receiving standard cardiac rehabilitation (Active Comparator): Consenting participants in this group will receive a standard cardiac rehabilitation protocol.
  Interventions: Other: Group A: Patients with FHP receiving standard cardiac rehabilitation
- Group B: Patients with FHP receiving standard cardiac rehabilitation + therapeutic exercises (Experimental): The participants who give consent will receive standard cardiac rehabilitation protocol (as Group A) with therapeutic exercise in the intervention group.
  Interventions: Other: Group B: Patients with FHP receiving standard cardiac rehabilitation + therapeutic exercises
- Group C: Patients without FHP receiving standard cardiac rehabilitation (Active Comparator): The participants without forward head posture will be included in this group and will receive same standard cardiac rehabilitation as the participants in group A.
  Interventions: Other: Group C: Patients without FHP receiving standard cardiac rehabilitation

INTERVENTIONS:
Other: Group A: Patients with FHP receiving standard cardiac rehabilitation — Consenting participants in this group will receive a standard cardiac rehabilitation protocol that includes preoperative education and post-operative exercises, chest physiotherapy, functional mobility and care. Phase 1 begins after the patient has been considered clinically compensated due to the optimization of the clinical treatment and/or the use of an interventional procedure. In this phase, a combination of low-intensity physical exercise (that includes range of motion exercises for upper & lower extremities + progressive mobilization from sitting on bedside to walking short distance and up to stair climbing), incentive spirometry exercise, percussions, breathing exercises and effective coughing exercises.
  Arms: Group A: Patients with FHP receiving standard cardiac rehabilitation
Other: Group B: Patients with FHP receiving standard cardiac rehabilitation + therapeutic exercises — The participants who give consent will receive standard cardiac rehabilitation protocol (as Group A) with therapeutic exercise in the intervention group.
  Therapeutic exercises will be delivered to the participant by treating physiotherapist in physical, verbal and written formats as individualized sessions on the ward 4 weeks before the surgery and keep him doing exercises under supervision while staying in the ward before surgery. A log will be provided to measure performance to ensure program compliance. After discharge from the hospital, the patient will continue exercises at home as performed and guided physically by the therapist and also in the exercises manual and flyer given to the patient. Patients will be instructed to follow therapeutic exercise for 4 weeks pre-operatively and 4 weeks postoperatively after discharge from the hospital.
  Arms: Group B: Patients with FHP receiving standard cardiac rehabilitation + therapeutic exercises
Other: Group C: Patients without FHP receiving standard cardiac rehabilitation — The participants without forward head posture will be included in this group and will receive same standard cardiac rehabilitation as the participants in group A.
  Arms: Group C: Patients without FHP receiving standard cardiac rehabilitation

SUMMARY:
Comparison of open heart surgery patients with forward head posture with and without perioperative therapeutic exercise on craniovertebral angle, pulmonary function, balance and quality of life

DETAILED DESCRIPTION:
Open heart surgery is at high risk of postoperative complications including pulmonary disorders, balance dysfunction and affects quality of life. These complications contribute to morbidity and mortality and increase hospitalization stay and its associated costs. The high prevalence of forward head posture (FHP) in the community is also associated with stated complications like pulmonary disorders, balance dysfunction and affecting quality of life. This close association of these complications in a person with forward head posture undergoing open heart surgery may further heighten the risks. The aim of this study is to evaluate the effects of therapeutic exercises on craniovertebral angle, pulmonary disorders, static and dynamic balance and quality of life in open heart surgery patient having forward head posture. This study will be a prospective, parallel-group, allocation concealment, randomized control, patient and assessor blind trial. Patients (n=53) who undergo open heart surgery via median sternotomy with forward head posture will be recruited from a cardiac hospital. Participants will be divided into three groups. Participants with FHP will be randomized into two groups; 1) patients with FHP will receive standard cardiac rehab protocol, 2) patients with FHP will receive standard cardiac rehab protocol with therapeutic exercise for forward head posture, and 3) participants without FHP will receive standard cardiac rehabilitation. The intervention group will receive a combination of stretching and strengthening exercises (including sternocleidomastoid stretch, pectoralis stretch, the supine chin tuck, and scapular retraction) for forward head posture with standard cardiac rehabilitation. The outcome measures will be craniovertebral angle, pulmonary parameters, neck disability index, functional difficulties questionnaire, single-leg stance test, forward reach test, health-related quality of life (SF-36), and Tampa scale for kinesiophobia. Repeated measures analysis of variance will be taken to test the hypothesis and to evaluate the change from baseline (4 weeks before surgery) to one day before surgery, after surgery before discharge and 4 weeks after discharge from the hospital in the intervention group compared with the standard-care group.

ELIGIBILITY:
Inclusion Criteria:

* Craniovertebral angle < 50 degrees (included in Group A & B), Craniovertebral angle ≥ 50 degree (included in Group C)
* First elective coronary artery bypass graft surgery, valve replacement, or both through a median sternotomy
* Extubated within 6 hours after surgery

Exclusion Criteria:

* Subjects with a history of surgery or any diagnosed pathology or clinical deformity or any musculoskeletal injury within the last six months to the spine or thorax or shoulder or lower extremity
* Any comorbid lung disease
* Patients having angina pectoris while doing therapeutic exercises
* Neurological dis¬orders, neuromuscular disorders, psychiatric, dizziness and blurred vision
* Inability to stand or walk independently
* Leg length discrepancy
* Have been reoperated on/ History of previous cardiac surgery
* Postoperative cardiac dysfunction, hemodynamically unstable, ventilator dependent
* Emergency cardiac surgery
* A length of stay in the intensive care unit for 5 days or more due to medical reasons after cardiac surgery
* Postoperative wound infections or sternal instability as diagnosed by medical staff

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | Baseline to nine weeks
  For measuring the angle, the reflective markers will be placed on the tragus of the ear and spinous process of the C7. The participant will be asked to stand and maintain her usual upright posture with her arms resting at the sides, and looking straight ahead. The photos will be captured by a digital camera. The camera will be positioned on a tripod 50 cm away from the participant. The axis of the lens of the camera will be placed orthogonal to the sagittal plane of the participant at the level of the shoulder. The photos will be taken repeatedly so that the participant was not exactly aware of the actual time of photography. The craniovertebral angle will be calculated by image. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Forced Vital Capacity (FVC) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Forced Expired Volume in one second (FEV1) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Forced Expired Volume in one second/Forced Vital Capacity (FEV1/FVC) ratio | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Peak expiratory flow (PEF) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
25% of the Force Expiratory Flow (FEF25) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
75% of the Force Expiratory Flow (FEF75) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Average flow between 25% and 75% of the Force Expiratory Flow (FEF25-75) | Baseline to nine weeks
  Spirometry is the term for basic lung function tests that measure the amount of air exhaled and inhaled. There are three basic related measurements: volume, time, and flow. Spirometry is objective, non-invasive, sensitive to early changes and reproducible. With the availability of portable measuring devices, it can be performed almost anywhere and by anyone with the right training. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Standing balance | Baseline to nine weeks
  The Single Leg Stance Test (SLST) is used to assess static balance performance which requires the participant to stand barefoot on their right or left leg (donor's leg) and hold the contralateral leg in approximately 45 degrees of hip flexion and 90 degrees of knee flexion. They are instructed to cross their arms over the chest. The assessor uses a digital chronometer to measure the amount of time patients are able to stand on a single limb. The test ends when the patient's legs touch each other, the non-stance leg touches the floor, or the arms move from the starting position. This process is repeated three times with eyes open and three times with eyes closed. A two-minute rest period between attempts is considered to prevent fatigue. The average of the three trials is calculated separately. The participants will be assessed at baseline, one day before surgery (±1 day) and 4 weeks post-discharge (±3 days).
Dynamic balance | Baseline to nine weeks
  The Functional Reach Test (FRT) is widely used as a dynamic measure of balance and is a reliable measure of balance for clinical assessment of instability. Participants are asked to stand with their dominant side adjacent to a wall and raise their arm to shoulder height. They are then asked to reach out as far forward as possible while maintaining a firm base of support. A tape measure is attached horizontally to the wall, and the maximum reach distance is recorded as the farthest point of the third metacarpophalangeal joint from the initial (standing) position. In other words, the measures the maximum distance the participants can reach forward from a standing static position. Three trials are performed and the mean value is recorded. The participants will be assessed at baseline, one day before surgery (±1 day) and 4 weeks post-discharge (±3 days).
Disability | Baseline to nine weeks
  Howard Vernon developed the Neck Disability Index (NDI) in 1989. The Neck Disability Index is now a standard tool to measure self-reported disability due to neck pain. This tool has 10 items and each score from 0 to 5. 50 is the maximum score. To get a percentage score, the score obtained is multiplied by two. The average of all other items is then added to the completed items, if a respondent will not answer one or other question,. NDI is a commonly used tool to measure disability in individuals with forward head posture. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Functional status | Baseline to nine weeks
  The Functional Difficulties Questionnaire measures the functional status of patients following cardiac surgery, with special emphasis on upper extremity and trunk function in patients following median sternotomy. The questionnaire asks patients to rate the difficulty they would experience performing a series of 13 functional upper extremity and trunk tasks. Specifically, patients are required to place a mark along a 10-cm line, with anchors to the left and right of the line, respectively indicating 'no difficulty' and 'maximum difficulty'. For the activities that participants cannot complete when completing the questionnaire, they are required to recall they performed the tasks last time. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Health related Quality of life | Baseline to nine weeks
  Health related quality of life is assessed by SF-36, a common measure used to assess eight domains including physical functioning, role physical functioning, role emotional functioning, mental health, vitality, social functioning, bodily pain and general health. All scale or single-item measurements range in score from 0 to 100 and are managed by interview. The raw subscale scores are converted to 'norm-based' scores using published algorithms. Norm-based total physical and mental component scores are calculated from the raw subscale scores, with higher scores indicating better quality of life. A higher score in the SF-36 subdomains is associated with a high level of functioning and higher quality of life. The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).
Pain-related fear beliefs | Baseline to nine weeks
  The TSK-11 is a widely used tool to measure pain-related fears related to movement and re-injury. It is an adaptation of the original 17-item instrument designed to assess fear of movement or re-injury excluding the 4 original reverse-scored items that were found to have small item-to-total score correlations. The adapted score is an 11-item tool that asks respondents to rate each item on a 4-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The TSK-11 is a reliable and valid measure of fear of movement or re-injury in patients with chronic pain. It has internal consistency, reliability and convergent validity with a Cronbach's α of 0.80 for the total score (Woby et al., 2005). The participants will be assessed at baseline, one day before surgery (±1 day), after surgery before discharge (7th postoperative day) (±1 day) and 4 weeks post-discharge (±3 days).

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, PhD scholar, Principal Investigator — Tehran University of Medical Sciences, Iran; Behrouz Attarbashi Moghadam, PhD, Study Chair — Tehran University of Medical Sciences, Iran; Azadeh Shadmehr, PhD, Study Chair — Tehran University of Medical Sciences, Iran
Locations (1):
- Rawalpindi Institute of Cardiology, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No